CLINICAL TRIAL: NCT03898713
Title: Assessment of Intellectual Abilities for Subjects With Velopharyngeal Incompetence and Their Impact on Speech Intelligibility
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeinab Abdel Ghani Abdel Hameed Mohamed, principle investigator at phoniatric department, Assiut University
Other Study IDs: IQ In VPI patients
Record Dates: First submitted 2019-03-24; First posted 2019-04-02 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Velopharyngeal Incompetence Due to Cleft Palate
Keywords: IQ; Speech; VPI
MeSH Terms: conditions — Speech

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Intelligence quotient — intelligence quotient (IQ) is a total score derived from several standardized tests designed to assess human intelligence

SUMMARY:
To Assess effect of intelligence on speech production on subjects with velopharyngeal incompetence Search if there is any relation between congenital Velopharyngeal incompetence and decrease IQ of patients

DETAILED DESCRIPTION:
Speech production is a complex process by which thoughts are generated into spoken utterances. Production involves the selection of appropriate words and the appropriate form of those words from the lexicon and morphology, and the organization of those words through the syntax. Then, the phonetic properties of the words are retrieved and the sentence is uttered through the articulations associated with those phonetic properties.

The term intelligibility refers to 'speech clarity' or the proportion of a speaker's output that a listener can readily understand.

Velopharyngeal Incompetence (VPI) refers to any situation in which an individual is unable to completely close the nasal airway during speech. The velopharyngeal mechanism is comprised of a complex group of structures that act in unison to control airflow through the nose and mouth by elevation of the soft palate and constriction of both the lateral and posterior pharyngeal walls. Any disruption in this mechanism may result in abnormal, poorly intelligible speech. VPI can manifest as hypernasality, nasal emission, decreased vocal intensity, and/or facial grimacing.

Intellectual ability refers to the skills required to think critically, see connections between disciplines and problem solve in new or changing situations. Memory, creative problem solving and vocabulary also contribute to the level of an individual's intellectual ability.

Orofacial clefts (OFCs) are frequently occurring human birth defects that have a complex, multifactorial etiology. Though structural orofacial defects are often surgically corrected during infancy and early childhood, OFC patient cohorts are at high risk for neurobehavioral problems including learning disability, impaired language function, psychosocial adjustment issues, and persistently reduced academic achievement.

ELIGIBILITY:
Inclusion Criteria:

* children with cleft lip and palate primary or secondary repaired
* Velopharyngeal incompetence due to any cause especially short palate and deep pharynx
* children above 3 years

Exclusion Criteria:

* Hearing impairment
* Neurological disease
* ADHD

Ages: 3 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients will be collected randomly for one year from phoniatric department at Assiut university Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Auditory perceptual assessment | Baseline
  Auditory-perceptual evaluation is the most commonly used clinical voice assessment method, and is often considered a gold standard for documentation of voice disorders.
IQ test | Baseline
  Assess IQ level of patients by standford binet version 4. An intelligence quotient (IQ) is a total score derived from several standardized tests designed to assess human intelligence.
  This is to search if there is any relation between IQ level and VPI and effect on speech intelligability

REFERENCES:
- [Background] Levelt WJ. Models of word production. Trends Cogn Sci. 1999 Jun;3(6):223-232. doi: 10.1016/s1364-6613(99)01319-4. PMID 10354575
- [Background] Robin NH, Baty H, Franklin J, Guyton FC, Mann J, Woolley AL, Waite PD, Grant J. The multidisciplinary evaluation and management of cleft lip and palate. South Med J. 2006 Oct;99(10):1111-20. doi: 10.1097/01.smj.0000209093.78617.3a. PMID 17100032
- [Background] Waitzman NJ, Romano PS, Scheffler RM. Estimates of the economic costs of birth defects. Inquiry. 1994 Summer;31(2):188-205. PMID 8021024
- See also: Related Info — https://www.nature.com/articles/mp201185